CLINICAL TRIAL: NCT04132856
Title: Mapping Psychosocial Screening to Services for Children With Cancer: Feasibility and Pilot Study
Brief Title: Mapping Psychosocial Screening to Services for Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Maru Barrera, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 1000056445
Record Dates: First submitted 2019-10-10; First posted 2019-10-21 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Cancer
Keywords: pediatric; oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The Intervention group will receive the services of the Psychosocial Navigator (PSN) monthly for the full 12 months of the study. At baseline, the PSN will provide the health care providers (HCPs) and family with recommendations for mapping and triaging of resources to levels of psychosocial risk (PAT: Universal, Targeted, Clinical) and level of depression and anxiety (mild, moderate, and high mental health problems; as determined by the standardized norms for the measures). This information will be summarized in the Communication Summary Profile and shared with the treating team (oncologist, nurse, and Social Worker, core psychosocial staff involved in the child's care) and family within 48 hours of completion. The PSN will conduct follow-up psychosocial screenings on a monthly basis, using the Distress Thermometer for children and caregivers. Results of the monthly assessments and recommended resources will also be communicated to the caregiver/parent and treating team of the youth.
  Interventions: Other: Psychosocial Navigator; Other: Communication of Summary Profile
- Treatment as Usual Group (No Intervention): Current psychosocial care services will be accessible to Treatment as Usual Group (e.g., social work, child life, psychology, art and music therapy, and psychiatry).

INTERVENTIONS:
Other: Psychosocial Navigator — Services of psychosocial navigator
  Arms: Intervention Group
Other: Communication of Summary Profile — Both patient/caregiver dyad and HCPs will receive a summary of the PAT results and levels of depression and anxiety.
  Arms: Intervention Group

SUMMARY:
Children with cancer are vulnerable to symptoms of anxiety and depression. Although screening for psychosocial distress is a standard of care for children with cancer, there is a limited knowledge

DETAILED DESCRIPTION:
Background: Approximately 3 000 children and adolescents are diagnosed with cancer in Canada each year [Canadian Cancer Society]. Children with cancer experience higher rates of anxiety and depression symptoms relative to healthy controls [Pinquart & Shen, 2011], and a subgroup are vulnerable to marked levels of psychological distress [Kurtz & Abrams, 2011]. One standard for psychosocial care in pediatric cancer that is starting to be implemented across the United Stated and Canada is the systematic screening for psychosocial distress, using the Psychosocial Assessment Tool (PAT) [Kazak, Schneider, Didonato, Pai, 2015; Pai et al., 2008; Barrera et al., 2014; McCarthy et al., 2009; Sint Nicolaas et al., 2016]. However, a dearth of literature exists on how to bridge screening for psychosocial distress and the delivery of appropriate evidence-based mental health resources. The current study is a randomized controlled pilot intervention project which aims to test the feasibility and effects of introducing a psychosocial navigator who will coordinate the delivery of psychosocial resources to children with cancer and their families based on early screening and follow-up for psychosocial distress. Specific Objectives: 1) To determine the feasibility and utility of conducting psychosocial screening and providing an Enhanced Psychosocial Intervention (EPSI). 2) To examine the effects of EPSI, as compared to treatment as usual (TAU+), on the mental health, quality of life, coping, and social relationships of children with cancer. Methods: A randomized controlled feasibility intervention trial, with a TAU+ control group, will be conducted with newly diagnosed children with any type of cancer. Participants will be 10-18 years of age, medically suitable for participation, in active treatment, and the primary caregiver. Forty-eight child-caregiver dyads (24 in the intervention and 24 in the control group) will be enrolled. The EPSI will have two components: 1) Information about the psychosocial risk of the family and mental health of the child (e.g., depression) and 2) the Psychosocial Navigator (PSN) as resource for tailoring psychosocial resources to child-family distress, linking with the treating team. Measures of feasibility (recruitment, acceptability) will be documented throughout; initial screening using the PAT will be conducted 2-4 weeks post diagnosis (baseline); and using the distress thermometer, follow-up will be done at specific periods depending on the disease (leukemia/lymphoma, solid tumors, brain tumors). The primary psychosocial outcome (depression), and secondary outcomes (post-traumatic stress, pain, fatigue, coping, sleep quality, time and financial cost, social support and quality of life) will be completed at baseline and 12 months later. Descriptive statistics (frequency and percentage rates) will be provided for feasibility measures and PAT psychosocial risk categories. Means, standard deviations, and ranges will be provided for the primary and secondary outcomes. Preliminary analyses of group comparisons will also be performed via independent t tests and chi square tests. Further, analyses of covariance (ANCOVAs) will be conducted on the primary and secondary outcomes to test group differences at post-test while controlling for pretest scores.

Significance: The proposed intervention project will assess and address the psychosocial needs of newly diagnosed pediatric cancer patients and families. This intervention aims to improve the triaging of resources and enhance the effectiveness of psychosocial intervention for children with cancer. The enhanced intervention is expected to improve children's and adolescents' coping with disease-related stressors such as pain and uncertainty, improve their mood, and enhance social engagement with peers.

ELIGIBILITY:
Inclusion Criteria:

* Between 10 and 18 years of age
* Clinical diagnosis of cancer
* Less than 4 weeks since diagnosis disclosure
* Primary caregiver must also consent to participation

Exclusion Criteria:

* Cancer diagnosis disclosed more than 4 weeks ago.
* Primary caregiver declines to participate

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Feasibility pertaining to recruitment | 12 months
  Rate of recruitment as measured by percentage of participants who consent to participation as compared to those who are eligible and do not consent
Feasibility pertaining to retention | 12 months
  Rates of completed questionnaires at all time points
Satisfaction with Enhanced Intervention as assessed by questionnaire at completion of study | 12 months
  5 - point likert scale satisfaction questionnaire with 6 questions pertaining to usefulness and overall satisfaction with the enhanced intervention. The minimum score is 6 (low satisfaction) and the maximum score is 30 (high satisfaction).
Satisfaction with Enhanced Intervention as assessed by semi-structured interview at completion of study | 12 months
  Semi-structured interview with 6 questions including "What were your expectations about being in this study?"; "Were your expectations of the study met?"; "Do you have any additional comments/suggestions for the study?"

SECONDARY OUTCOMES:
Distress | Change from baseline to 12 months
  Pediatric and Adult Distress Thermometer (self-report) measures participant distress on a visual analog scale of 1 to 10, with a score of 10 indicating high distress
Patient generic quality of life based on self report | Change from baseline to 12 months
  Pediatric Quality of Life - generic. (Child/teen self-report). Measures perceived quality of life of child with cancer based on self perception - on everyday items (for children who do not have cancer). Miinimum score is 0. Maximum score is 100. Higher score indicates better perceived quality of life.
Patient generic quality of life based on caregiver report | Change from baseline to 12 months
  Pediatric Quality of Life - generic. (Caregiver-report). Measures perceived quality of life of child with cancer based on caregiver perception - on everyday items (for children who do not have cancer). Miinimum score is 0. Maximum score is 100. Higher score indicates better perceived quality of life.
Patient quality of life as it relates to cancer, based on self-report | Change from baseline to 12 months
  Pediatric Quality of Life-Cancer (Child/teen self-report). Measures perceived quality of life of child with cancer based on self-perception. Miinimum score is 0. Maximum score is 100. Higher score indicates better perceived quality of life.
Patient quality of life as it relates to cancer, based on caregiver report | Change from baseline to 12 months
  Pediatric Quality of Life-Cancer (Caregiver report). Measures perceived quality of life of child with cancer based on caregiver perception. Miinimum score is 0. Maximum score is 100. Higher score indicates better perceived quality of life.
Patient anxiety and depression - child/teem self report | Change from baseline to 12 months
  Pediatric Index of Emotional Distress. Minimum score is 0. Maximum score is 42. Lower score indicates lower levels of anxiety and depression.
Patient anxiety (child/teen self-report) | Change from baseline to 12 months
  Patient-reported Outcomes Measurement Information System (PROMIS) - pediatric anxiety questionnaire - short form (child/teen self-report). Minimum score is 8. Maximum score is 40. Lower score indicates lower level of anxiety.
Patient depression (child/teen self-report) | Change from baseline to 12 months
  Patient-reported Outcomes Measurement Information System (PROMIS) - pediatric depression questionnaire - short form (child/teen self-report). Minimum score is 8. Maximum score is 40. Lower score indicates lower level of depression.
Caregiver post-traumatic stress related to child's cancer diagnosis | Change from baseline to 12 months
  Impact of Events scale - Revised (IES-R) (caregiver self-report). Mimimum score is 0. Maximum score is 88. Lower scores indicate lower levels of post-traumatic stress.
Patient post-traumatic stress related to own cancer diagnosis | Change from baseline to 12 months
  Impact of Events scale - Revised (IES-R) (child/teen self-report). Mimimum score is 0. Maximum score is 88. Lower scores indicate lower levels of post-traumatic stress.
Caregiver coping with stress of child's cancer diagnosis | Change from baseline to 12 months
  Responses to Stress Questionnaire - Cancer Version (caregiver self-report). Minimum score is 0. Maximum score is 1. A higher score indicates more engagement with active coping strategies.
Patient's own coping with stress of cancer diagnosis | Change from baseline to 12 months
  Response to Stress Questionnaire - Cancer Version (patient self-report). Minimum score is 0. Maximum score is 1. A higher score indicates more engagement with active coping strategies.
Psychosocial risk | Change from baseline to 12 months
  Psychosocial Assessment Tool (PAT) (caregiver report). Minimum score is 0. Maximum score is 3. Lower score indicates lower level of psychosocial risk.
Financial impact of pediatric cancer diagnosis and treatment on families. | Change from baseline to 12 months
  Financial burden questionnaire (caregiver report). Minimum score is 22. Maximum score is 88. Higher score indicates lower level of financial impact on families.
Caregiver depression | Change from baseline to 12 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Questionnaire (caregiver self-report). Minimum score is 6. Maximum score is 30. Lower scores indicate lower levels of depression.
Caregiver anxiety | Change from baseline to 12 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Questionnaire (caregiver self-report). Minimum score is 6. Maximum score is 30. Lower scores indicate lower levels of anxiety.

OTHER OUTCOMES:
Sleep duration and quality of sleep of patient and caregiver | Change from baseline to 12 months
  Pittsburgh Sleep Quality Index. (Caregiver and patient self-report). Minimum value is 0. Maximum value is 21. Lower scores indicate better sleep quality.
Caregiver emotional support | Change from baseline to 12 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Support Questionnaire (caregiver self-report). Minimum score is 6. Maximum score is 30. Higher scores indicate higher levels of emotional support.
Caregiver Fatigue | Change from baseline to 12 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Questionnaire (caregiver self-report). Minimum score is 6. Maximum score is 30. Lower scores indicate lower levels of fatigue
Patient Peer Relationships | Change from baseline to 12 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) Perceived Quality of Peer Relationships (child/teen self-report). Minimum score is 8. Maximum score is 40. Higher scores indicate higher levels of perceived peer relationship quality.
Patient Fatigue | Change from baseline to 12 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Questionnaire (child/teen self-report). Minimum score is 10. Maximum score is 50. Lower scores indicate lower levels of fatigue.
Patient emotional support | Change from baseline to 12 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Support Questionnaire (child/teen self-report). Minimum score is 7. Maximum score is 35. Higher scores indicate higher levels of emotional support.

CONTACTS AND LOCATIONS:
Overall Officials: Maru Barrera, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canadian Cancer Society's Advisory Committee on Cancer Statistics. Canadian Cancer Statistics 2015. Toronto, ON: Canadian Cancer Society; 2015.
- [Background] Pinquart M, Shen Y. Behavior problems in children and adolescents with chronic physical illness: a meta-analysis. J Pediatr Psychol. 2011 Oct;36(9):1003-16. doi: 10.1093/jpepsy/jsr042. Epub 2011 Aug 1. PMID 21810623
- [Background] Kurtz BP, Abrams AN. Psychiatric aspects of pediatric cancer. Pediatr Clin North Am. 2011 Aug;58(4):1003-23, xii. doi: 10.1016/j.pcl.2011.06.009. PMID 21855719
- [Background] Kazak AE, Schneider S, Didonato S, Pai AL. Family psychosocial risk screening guided by the Pediatric Psychosocial Preventative Health Model (PPPHM) using the Psychosocial Assessment Tool (PAT). Acta Oncol. 2015 May;54(5):574-80. doi: 10.3109/0284186X.2014.995774. Epub 2015 Mar 9. PMID 25752970
- [Background] Pai AL, Patino-Fernandez AM, McSherry M, Beele D, Alderfer MA, Reilly AT, Hwang WT, Kazak AE. The Psychosocial Assessment Tool (PAT2.0): psychometric properties of a screener for psychosocial distress in families of children newly diagnosed with cancer. J Pediatr Psychol. 2008 Jan-Feb;33(1):50-62. doi: 10.1093/jpepsy/jsm053. Epub 2007 Jul 3. PMID 17609228
- [Background] Barrera M, Hancock K, Rokeach A, Cataudella D, Atenafu E, Johnston D, Punnett A, Nathan PC, Bartels U, Silva M, Cassidy M, Jansen P, Shama W, Greenberg C. External validity and reliability of the Psychosocial Assessment Tool (PAT) among Canadian parents of children newly diagnosed with cancer. Pediatr Blood Cancer. 2014 Jan;61(1):165-70. doi: 10.1002/pbc.24774. Epub 2013 Sep 17. PMID 24106172
- [Background] McCarthy MC, Clarke NE, Vance A, Ashley DM, Heath JA, Anderson VA. Measuring psychosocial risk in families caring for a child with cancer: the Psychosocial Assessment Tool (PAT2.0). Pediatr Blood Cancer. 2009 Jul;53(1):78-83. doi: 10.1002/pbc.22007. PMID 19343796
- [Background] Sint Nicolaas SM, Schepers SA, Hoogerbrugge PM, Caron HN, Kaspers GJ, van den Heuvel-Eibrink MM, Grootenhuis MA, Verhaak CM. Screening for Psychosocial Risk in Dutch Families of a Child With Cancer: Reliability, Validity, and Usability of the Psychosocial Assessment Tool. J Pediatr Psychol. 2016 Aug;41(7):810-9. doi: 10.1093/jpepsy/jsv119. Epub 2015 Dec 29. PMID 26715054
- [Derived] Desjardins L, Hancock K, Szatmari P, Alexander S, Shama W, De Souza C, Mills D, Abla O, Barrera M. Protocol for mapping psychosocial screening to resources in pediatric oncology: a pilot randomized controlled trial. Pilot Feasibility Stud. 2021 Jul 17;7(1):143. doi: 10.1186/s40814-021-00878-0. PMID 34274016